CLINICAL TRIAL: NCT01563172
Title: A Study to Measure the Effect of Dentifrice Usage Regime on Delivery and Efficacy of Fluoride Using an In Situ Caries Model
Brief Title: Effect of Dentifrice Usage Regime on Delivery and Efficacy of Fluoride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: T3158587
Record Dates: First submitted 2012-02-16; First posted 2012-03-26 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Sodium Fluoride; Silicon Dioxide; carboxypolymethylene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Experimental dentifrice 0.5g, 45 seconds brushing group (Experimental): Participants brush twice a daily for 45 seconds with experimental dentifrice.
  Interventions: Drug: Sodium fluoride / silica and carbopol, 0.5g; Other: Fluoride free dentifrice
- Experimental dentifrice 1.5g, 45 seconds brushing group (Experimental): Participants brush twice a daily for 45 seconds with experimental dentifrice.
  Interventions: Drug: Sodium fluoride / silica and carbopol, 1.5g; Other: Fluoride free dentifrice
- Experimental dentifrice 0.5g, 2 minutes brushing group (Experimental): Participants brush twice a daily for 2 minutes with experimental dentifrice.
  Interventions: Drug: Sodium fluoride / silica and carbopol, 0.5g; Other: Fluoride free dentifrice
- Experimental dentifrice 1.5g, 2 minutes brushing group (Experimental): Participants brush twice a daily for 2 minutes with experimental dentifrice.
  Interventions: Drug: Sodium fluoride / silica and carbopol, 1.5g; Other: Fluoride free dentifrice
- Contol group (Active Comparator): Participants brush twice a daily for 2 minutes with controll dentifrice.
  Interventions: Drug: Sodium fluoride / silica and carbopol, 1.5g; Other: Fluoride free dentifrice

INTERVENTIONS:
Drug: Sodium fluoride / silica and carbopol, 0.5g — Dentifrice containing 1150 parts per million (ppm) fluoride as sodium fluoride / silica and 0.4% carbopol
  Arms: Experimental dentifrice 0.5g, 2 minutes brushing group; Experimental dentifrice 0.5g, 45 seconds brushing group
Drug: Sodium fluoride / silica and carbopol, 1.5g — Dentifrice containing 1150 ppm fluoride as sodium fluoride / silica and 0.4% carbopol
  Arms: Experimental dentifrice 1.5g, 2 minutes brushing group; Experimental dentifrice 1.5g, 45 seconds brushing group
Drug: Sodium fluoride / silica and carbopol, 1.5g — Dentifrice containing 250 ppm fluoride as sodium fluoride / silica and 0.4% carbopol
  Arms: Contol group
Other: Fluoride free dentifrice — A non fluoride dentifrice was given to participants of each arm at washout period

SUMMARY:
This study will evaluate and compare the effect of the amount of toothpaste used and brushing time on enamel strengthening (percent of surface microhardness recovery, % SMHR) and enamel fluoride uptake (EFU).

ELIGIBILITY:
Inclusion Criteria:

General and Dental Health

* Good general and dental health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral examination
* Have no current active caries or periodontal disease that may compromise the study or the health of the subjects
* Residency: Currently living in the Indianapolis, Indiana area

Dentures:

* Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accommodate two enamel specimens (required dimensions 12 mm x 7 mm)
* Willing to have their denture modified to accommodate enamel test specimens and willing and capable of wearing their removable mandibular partial dentures 24 hours per day during the experimental periods
* All restorations in a good state of repair
* Salivary Flow: Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/minute; gum base stimulated whole saliva flow rate ≥ 0.8 mL/minute)

Exclusion Criteria:

* Antibiotics: Use of antibiotics two weeks prior to a treatment visit or anticipated use during the study treatment periods
* Study Scale Use: Subjects unable to measure product weights accurately using the assigned study scale as determined by the study staff (as demonstrated on or before Visit 4)
* A member of the site study staff who is directly working on the project or living in that staff's household
* Any employee of any toothpaste manufacturer or their spouse or family member

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

REFERENCES:
- [Result] https://clinicaltrials.gov/ct2/show/results/NCT01563172?term=T3158587&rank=1
- [Derived] Creeth JE, Kelly SA, Gonzalez-Cabezas C, Karwal R, Martinez-Mier EA, Lynch RJM, Bosma ML, Zero DT. Effect of toothbrushing duration and dentifrice quantity on enamel remineralisation: An in situ randomized clinical trial. J Dent. 2016 Dec;55:61-67. doi: 10.1016/j.jdent.2016.10.003. Epub 2016 Oct 4. PMID 27717756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 center in the USA.
Pre-assignment Details: Total of 74 participants were screened for the study, out of which 65 participants were randomized in the study. Nine participants were screen failures.
Groups:
- Overall: This was a five arm cross-over study. Five arms were divided according to the different treatment regimens, the participants were received all the following treatment regimens during the study: 1. Experimental dentifrice 0.5 grams (g) for 45 seconds, 2. Experimental dentifrice 0.5g for 2 minutes, 3. Experimental dentifrice 1.5g for 45 seconds, 4. Experimental dentifrice 1.5g for 2 minutes, and 5. Control dentifrice 1.5g for 2 minutes only.
Period: Overall Study
Arm/Group | Overall
Started | 65
Experimental Dentifrice 0.5g/2 Min | 59
Experimental Dentifrice 0.5g/45 Sec | 59
Experimental Dentifrice 1.5g/ 2min | 58
Experimental Dentifrice 1.5g/ 45 Sec | 58
Control Dentifrice | 60
Completed | 52
Not Completed | 13
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 2
Not completed — Other (Protocol deviation) | 5
Not completed — Other (Not specified) | 1

BASELINE CHARACTERISTICS:
Population: Safety population: The overall Safety Population included all the participants who were randomized and used at least one of the treatment dentifrices during the study and had at least one safety assessment (e.g. assessment of adverse events [AEs] or had an oral soft tissue examination) after using the treatment dentifrices.
Arm/Group | Overall
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 28
  Black | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Micro Hardness Recovery (% SMH), of Brushing for 2 Minutes Versus (vs.) Brushing for 45 Seconds With 1.5g of Experimental Dentifrice.
Description: SMH recovery test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH recovery was performed in-vitro and determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents re-hardening of enamel surface. % SMH recovery was calculated from indentation length (micrometer [μm]) of sound enamel specimen at baseline (B), indentation length (μm) after in vitro demineralization (D1), indentation length (μm) after intra-oral exposure (R): [D1-R/D1-B] ×100.
Time Frame: At Baseline and at Day 14
Population: Per Protocol (PP) population: Included all randomized participants who had no major protocol deviations that were felt by the investigator to have affected the assessment of efficacy for all treatments.
Measure: Least Squares Mean (Standard Error); unit: % SMH
Groups:
- Experimental Dentifrice 1.5g, 2 Minutes Brushing Group: Participants in this arm brushed their teeth twice a daily (morning and evening) for 2 minutes with 1.5g dose of experimental dentifrice.
- Experimental Dentifrice 1.5g, 45 Seconds Brushing Group: Participants in this arm brushed their teeth twice a daily (morning and evening) for 45 seconds with 1.5g dose of experimental dentifrice.
Arm/Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group | Experimental Dentifrice 1.5g, 45 Seconds Brushing Group
Number analyzed (Participants) | 57 | 53
% SMH | 41.61 (2.244) | 34.66 (2.284)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1.5g, 2 Minutes Brushing Group vs Experimental Dentifrice 1.5g, 45 Seconds Brushing Group; Test type: Superiority or Other; p = 0.0008, ANOVA — Between Treatment p-Values based on the statistical model adjusting for treatment, study period, and participant (random effect); Least square (LS) mean difference = 6.95, 95% CI 2-sided [2.91 to 10.98] — LS Mean from Analysis of variance (ANOVA) with factors for treatment, study period, and participant (random effect). Difference is first named treatment minus second named treatment such that a positive difference favours the first named treatment

2. Secondary Outcome: Percentage Surface Micro Hardness (% SMH) Recovery , of Brushing for 2 Minutes vs. Brushing for 45 Seconds With 0.5g of Experimental Dentifrice.
Description: SMH recovery test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH recovery was performed in-vitro and determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents re-hardening of enamel surface. % SMH recovery was calculated from indentation length (μm) of sound enamel specimen at baseline (B), indentation length (μm) after in vitro demineralization (D1), indentation length (μm) after intra-oral exposure (R): [D1-R/D1-B] ×100.
Time Frame: At Baseline and at Day 14
Population: PP population included all randomized participants who had no major protocol deviations that were felt by the investigator to have affected the assessment of efficacy for all treatments.
Measure: Least Squares Mean (Standard Error); unit: % SMH
Groups:
- Experimental Dentifrice 0.5g, 2 Minutes Brushing Group: Participants in this arm brushed their teeth twice a daily (morning and evening) for 2 minutes with 0.5g dose of experimental dentifrice.
- Experimental Dentifrice 0.5g, 45 Seconds Brushing Group: Participants in this arm brushed their teeth twice a daily (morning and evening) for 45 seconds with 0.5g dose of experimental dentifrice.
Arm/Group | Experimental Dentifrice 0.5g, 2 Minutes Brushing Group | Experimental Dentifrice 0.5g, 45 Seconds Brushing Group
Number analyzed (Participants) | 58 | 55
% SMH | 30.75 (2.232) | 25.05 (2.266)
Statistical Analysis 1: Comparison: Experimental Dentifrice 0.5g, 2 Minutes Brushing Group vs Experimental Dentifrice 0.5g, 45 Seconds Brushing Group; Test type: Superiority or Other; p = 0.0049, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 5.70, 95% CI 2-sided [1.74 to 9.66] — LS Mean from ANOVA with factors for treatment, study period, and participant (random effect). Difference is first named treatment minus second named treatment such that a positive difference favours the first named treatment

3. Secondary Outcome: Percentage Surface Micro Hardness (% SMH) Recovery, of Brushing for 2 Minutes With 0.5g of Experimental Dentifrice vs. Brushing for 2 Minutes With 1.5g of Experimental Dentifrice.
Description: as for outcome 2
Time Frame: At Baseline and at Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: % SMH
Arm/Group | Experimental Dentifrice 0.5g, 2 Minutes Brushing Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group
Number analyzed (Participants) | 58 | 57
% SMH | 30.75 (2.232) | 41.61 (2.244)
Statistical Analysis 1: Comparison: Experimental Dentifrice 0.5g, 2 Minutes Brushing Group vs Experimental Dentifrice 1.5g, 2 Minutes Brushing Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -10.86, 95% CI 2-sided [-14.77 to -6.94] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage Surface Micro-hardness Recovery (% SMH), of Brushing for 45 Seconds With 0.5g of Experimental Dentifrice vs. Brushing for 45 Seconds With 1.5g of Experimental Dentifrice.
Description: as for outcome 2
Time Frame: At Baseline and at Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: % SMH
Arm/Group | Experimental Dentifrice 0.5g, 45 Seconds Brushing Group | Experimental Dentifrice 1.5g, 45 Seconds Brushing Group
Number analyzed (Participants) | 55 | 53
% SMH | 25.05 (2.266) | 34.66 (2.284)
Statistical Analysis 1: Comparison: Experimental Dentifrice 0.5g, 45 Seconds Brushing Group vs Experimental Dentifrice 1.5g, 45 Seconds Brushing Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -9.61, 95% CI 2-sided [-13.68 to -5.54] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percent Surface Micro-hardness (% SMH) Recovery, of Brushing for 2 Minutes With 1.5g of Experimental Dentifrice vs. Brushing for 2 Minutes With 1.5g of an Control Dentifrice.
Description: as for outcome 2
Time Frame: At Baseline and at Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: % SMH
Groups:
- Contol Group: Participants in this arm brushed their teeth twice a daily (morning and evening) for 2 minutes with 1.5g dose of control dentifrice.
Arm/Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group | Contol Group
Number analyzed (Participants) | 57 | 58
% SMH | 41.61 (2.244) | 26.23 (2.232)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1.5g, 2 Minutes Brushing Group vs Contol Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 15.38, 95% CI 2-sided [11.45 to 19.31] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Enamel Fluoride Uptake (EFU) After Brushing for 2 Minutes vs. Brushing for 45 Seconds With 1.5g of Experimental Dentifrice.
Description: EFU was measured by using micro-drill analysis of the enamel specimens carried out after 14 days of intra-oral exposure for each of the toothpaste treatments. The amount of fluoride-uptake by enamel was calculated based on the amount of fluoride divided by the area of the enamel cores.
Time Frame: At Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micrograms (μg)×F/centimeters(cm)2
Arm/Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group | Experimental Dentifrice 1.5g, 45 Seconds Brushing Group
Number analyzed (Participants) | 57 | 53
micrograms (μg)×F/centimeters(cm)2 | 2426.51 (103.802) | 1912.51 (106.620)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1.5g, 2 Minutes Brushing Group vs Experimental Dentifrice 1.5g, 45 Seconds Brushing Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 514.01, 95% CI 2-sided [283.02 to 744.99] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Enamel Fluoride Uptake (EFU) After Brushing for 2 Minutes vs. Brushing for 45 Seconds With 0.5g of Experimental Dentifrice.
Description: as for outcome 6
Time Frame: At Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μg×F/cm2
Arm/Group | Experimental Dentifrice 0.5g, 2 Minutes Brushing Group | Experimental Dentifrice 0.5g, 45 Seconds Brushing Group
Number analyzed (Participants) | 58 | 55
μg×F/cm2 | 1603.63 (103.018) | 1337.72 (105.260)
Statistical Analysis 1: Comparison: Experimental Dentifrice 0.5g, 2 Minutes Brushing Group vs Experimental Dentifrice 0.5g, 45 Seconds Brushing Group; Test type: Superiority or Other; p = 0.0218, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean difference = 265.92, 95% CI 2-sided [39.00 to 492.83] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Enamel Fluoride Uptake (EFU) After Brushing for 2 Minutes With 0.5g of Experimental Dentifrice vs. Brushing for 2 Minutes With 1.5g of Experimental Dentifrice.
Description: as for outcome 6
Time Frame: At Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μg×F/cm2
Arm/Group | Experimental Dentifrice 0.5g, 2 Minutes Brushing Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group
Number analyzed (Participants) | 58 | 57
μg×F/cm2 | 1603.63 (103.018) | 2426.51 (103.802)
Statistical Analysis 1: Comparison: Experimental Dentifrice 0.5g, 2 Minutes Brushing Group vs Experimental Dentifrice 1.5g, 2 Minutes Brushing Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -822.88, 95% CI 2-sided [-1047.34 to -598.42] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Enamel Fluoride Uptake (EFU) After Brushing for 45 Seconds With 0.5g of Experimental Dentifrice vs. Brushing for 45 Seconds With 1.5g of Experimental Dentifrice.
Description: as for outcome 6
Time Frame: At Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μg×F/cm2
Arm/Group | Experimental Dentifrice 0.5g, 45 Seconds Brushing Group | Experimental Dentifrice 1.5g, 45 Seconds Brushing Group
Number analyzed (Participants) | 55 | 53
μg×F/cm2 | 1337.72 (105.260) | 1912.51 (106.620)
Statistical Analysis 1: Comparison: Experimental Dentifrice 0.5g, 45 Seconds Brushing Group vs Experimental Dentifrice 1.5g, 45 Seconds Brushing Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -574.79, 95% CI 2-sided [-808.08 to -341.50] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Enamel Fluoride Uptake (EFU) After Brushing for 2 Minutes With 1.5g of Experimental Dentifrice vs. Brushing for 2 Minutes With 1.5g of Control Dentifrice.
Description: as for outcome 6
Time Frame: At Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μg×F/cm2
Arm/Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group | Contol Group
Number analyzed (Participants) | 57 | 58
μg×F/cm2 | 2426.51 (103.802) | 1132.18 (103.044)
Statistical Analysis 1: Comparison: Experimental Dentifrice 1.5g, 2 Minutes Brushing Group vs Contol Group; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1294.34, 95% CI 2-sided [1069.24 to 1519.43] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately 16 Weeks
Description: All non-oral Adverse events (AEs) were not coded, therefore all the non-oral AEs were reported under system order class (SOC) General disorder.
Groups:
- Contol Group: Participants in this arm brushed their teeth twice a daily (morning and evening) for 2 minutes with control dentifrice.
Arm/Group | Experimental Dentifrice 0.5g, 45 Seconds Brushing Group | Experimental Dentifrice 0.5g, 2 Minutes Brushing Group | Experimental Dentifrice 1.5g, 45 Seconds Brushing Group | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group | Contol Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/58 | 0/58 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/58 | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 11/59 | 8/59 | 12/58 | 10/58 | 10/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Dentifrice 0.5g, 45 Seconds Brushing Group (N=59) | Experimental Dentifrice 0.5g, 2 Minutes Brushing Group (N=59) | Experimental Dentifrice 1.5g, 45 Seconds Brushing Group (N=58) | Experimental Dentifrice 1.5g, 2 Minutes Brushing Group (N=58) | Contol Group (N=60)
Gingival mucosa imprint from teeth 28 and 29 (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Common cold (General disorders) | 3 | 2 | 3 | 2 | 1
Cellulitis lower right leg (General disorders) | 1 | 0 | 0 | 0 | 0
Sore throat left side (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sprained right ankle (General disorders) | 1 | 0 | 0 | 0 | 0
Sinus infection (General disorders) | 1 | 0 | 0 | 0 | 0
Kidneys infection (General disorders) | 1 | 0 | 0 | 0 | 0
Erythema anterior hard palate (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gout (General disorders) | 1 | 0 | 0 | 0 | 0
Gingival mucosa edentulous maxillary anterior ridge erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Swelling of right inside of mouth & lip caused by biting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Felt very tired (General disorders) | 0 | 1 | 0 | 0 | 0
Ulceration on gingival lingual 26 ~2mm (millimeter) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival mucosa cervical lingual area swollen with exudate (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Back pain from arthritis (General disorders) | 0 | 1 | 0 | 0 | 0
Gout flare-up (General disorders) | 0 | 1 | 0 | 0 | 0
Gingival mucosa erythema of right posterior edentulous ridge (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival mucosa erythema left posterior edentulous ridge (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (General disorders) | 0 | 0 | 1 | 1 | 0
Boil on vaginal area (General disorders) | 0 | 0 | 1 | 0 | 0
White coating on tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest pains (General disorders) | 0 | 0 | 1 | 0 | 0
Worsening of acid reflux (General disorders) | 0 | 0 | 1 | 0 | 0
Mycosis fungoides of the skin (General disorders) | 0 | 0 | 1 | 0 | 0
Sore area on ridge area #22 from partial (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Submandibular area small ulcer not painful (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Seasonal allergies (General disorders) | 0 | 0 | 1 | 0 | 0
Lower back pain (General disorders) | 0 | 0 | 0 | 1 | 0
Diverticulitis (General disorders) | 0 | 0 | 0 | 1 | 0
Sinus drainage (General disorders) | 0 | 0 | 0 | 1 | 0
Erythema facial (General disorders) | 0 | 0 | 0 | 1 | 0
Brown coating on tongue (General disorders) | 0 | 0 | 0 | 1 | 1
Gingival mucosa erythema lingual tooth 23 (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dizziness and vomiting (General disorders) | 0 | 0 | 0 | 1 | 0
Broke right hip (right intertrochanteric hip fracture) (General disorders) | 0 | 0 | 0 | 1 | 0
Worsening of arthritis (General disorders) | 0 | 0 | 0 | 0 | 1
Thermal burn anterior hard palate (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Infected tooth 10 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Left eye swollen and red beneath eye (General disorders) | 0 | 0 | 0 | 0 | 1
Stomach virus (General disorders) | 0 | 0 | 0 | 0 | 1
Labial mucosa chapped lips upper & lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Crown come off tooth 9 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Right shoulder pain (General disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.